CLINICAL TRIAL: NCT06507501
Title: Effects of Exercise Training with Blood Flow Restriction on Lower Extremity Muscle Strength, Balance, Functional and Cognitive Performance in Healthy Individuals
Brief Title: Effects of Exercise Training with Blood Flow Restriction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Onur Turan, Research Assisstant, Atlas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Onur1
Record Dates: First submitted 2024-06-27; First posted 2024-07-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Blood Flow Restriction Exercise Training; Muscle Strength; Balance; Functional Performance; Cognitive Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Flow Restriction Exercise Training (BFRT) (Experimental): Exercises will be performed under the supervision of a researcher physiotherapist, at low intensity and progressively, under blood flow restriction for 6 weeks, 2 days a week, for a total of 12 exercise sessions. The 1 MT method will be used to determine the amount of resistance in strengthening exercises.
  Blood flow restriction will be made by wearing a pneumatic tourniquet from the proximal thigh, within a safe pressure range specific to each individual.
  Blood flow restriction United States Food and Drug Administration Using the (FDA) approved H+Cuff device, it will be applied for 20 minutes, with a 1-minute break between exercises. The cuff pressure will be maintained during the rest period, and after the application, individuals will rest for 15 minutes to ensure reperfusion and other exercises will continue.
  Interventions: Other: Low Load Blood Flow Restriction Exercise Training (LL-BFRE)
- Conventional Exercise Training (Experimental): Participants who will be included in the conventional exercise group will apply the same exercise program as the participants in the blood flow-restricted exercise group, without blood flow restriction, for 6 weeks, 2 days a week, in a total of 12 sessions, at medium-high intensity.
  Interventions: Other: High Load Resistive Exercise Training (HL-RE)

INTERVENTIONS:
Other: Low Load Blood Flow Restriction Exercise Training (LL-BFRE) — Blood Flow Restriction exercise training, also known as occlusion training or KAATSU training, is a contemporary exercise training method based on partially restricting arterial and venous blood flow for short periods.
  Arms: Blood Flow Restriction Exercise Training (BFRT)
Other: High Load Resistive Exercise Training (HL-RE) — HL-RE is a conventional, well known exercise method to enhance muscle strength and improve physical performance. It's performed by using resistance bands or weights applying on the extremity.
  Arms: Conventional Exercise Training

SUMMARY:
In this study, it was aimed to compare the effects of low load blood flow restriction exercise (LL-BFRE) training versus high load resistance exercise (HL-RE) training in healthy young individuals on the parameters of lower extremity muscle strength, dynamic and static postural balance, functional performance and cognitive performance.

DETAILED DESCRIPTION:
In this randomized controlled study, there will be two study group. Study group 1 will recieve low load blood flow restriction exercise training and Study group 2 will recieve high load resistance exercise training for 6 weeks, 2 exercise sessions weekly.

At baseline assessment, individuals who met the inclusion criteria, informed by the researcher and accept the participate in the study, researcher will record the participants' sociodemographic and physical informations and then, asess the lower extremity muscle strength with Hand-held digital dynamometer, dynamic postural balance with Y-Balance Test-Lower Quarter, static postural balance with Single Leg Stance Test (Eyes open/closed condition), functional performance with 6-Minute Walking Test and cognitive performance with Stroop Word and Colour Test and Trail Making Test.

At the end of the 6 week exercise training all participants will undergo the same assessments.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* Being between the ages of 18-30.

Exclusion Criteria:

* Presence of any painful condition or pathology involving the lower extremity and lumbar spine and the presence of a surgical history,
* Presence of serious malalignment and deformity affecting the lower extremity,
* Presence of neuromuscular and metabolic disease,
* Presence of any disease affecting lower extremity circulation,
* Having a history of deep vein thrombosis and the presence of peripheral vascular disease,
* Presence of endothelial dysfunction (ED) and any disease that may cause ED,
* Presence of active infection, cancer and having received radiotherapy / chemotherapy,
* Continuous use of anticoagulant medication,
* Having had COVID-19 in the last 3 months or having long COVID syndrome,
* Presence of a cognitive or mental disorder that would disability to participate in the study,
* Disruption of exercise program 3 times in a row

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Baseline to 6 weeks after exercise training
  Knee extansor and flexor muscle strength will be measured by using Hoggan Scientific; MicroFET2 brand hand-held dynamometer.
Dynamic Balance | Baseline to 6 weeks after exercise training
  Dynamic balance will be assessed by using Y-Balance Test Lower Extremity.
Static Balance | Baseline to 6 weeks after exercise training
  Static balance will be assessed by using Single Leg Stance Test with eyes open and closed.

SECONDARY OUTCOMES:
Funtional Performance | Baseline to 6 weeks after exercise training
  Functional performance will be assessed by using 6 Minute Walk Test.
Funtional Performance | Baseline to 6 weeks after exercise training
  Functional performance will be assessed by using Single Leg Hop Test.
Cognitive Performance | Baseline to 6 weeks after exercise training
  Cognitive performance will be assessed by using Trail Making Test.
Cognitive Performance | Baseline to 6 weeks after exercise training
  Cognitive performance will be assessed by using Stroop Colour and Word Test.

OTHER OUTCOMES:
Sociodemographic Information | Baseline
  Age (years), gender, education level, smoking & alcohol habits, whether they have a chronic disease, whether they use any medication, and exercise habits of the individuals participating in the study will be recorded.
Physical Assessment | Baseline
  Height (cm), body weight (kg) and body mass index (BMI) (kg/m2) will be measured. Height will be measure via stadiometer, body weight will be measure via weighing device and BMI will be calculated using with the formula "weight/height (m)2".

CONTACTS AND LOCATIONS:
Overall Officials: Onur Turan, Bachelor's, Principal Investigator — Atlas University
Locations (1):
- Onur Turan, Istanbul, Kağıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No